CLINICAL TRIAL: NCT06222632
Title: Cardioprotective and Mental Health Benefits of the Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Diet Combined With Forest Bathing (FB) Among Adults With Elevated Blood Cholesterol: A Randomized Controlled Trial
Brief Title: Cardioprotective and Mental Health Benefits of the MIND Diet Combined With Forest Bathing
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tung Wah College (Other)
Responsible Party: Principal Investigator, Katherine Yau, Assistant Professor, Tung Wah College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REC2023164; UGC/FDS17/H01/23 (Other Grant/Funding Number: University Grants Committee_Faculty development scheme)
Record Dates: First submitted 2023-12-26; First posted 2024-01-25 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Elevated LDL Cholesterol
Keywords: MIND diet; Forest bathing; LDL cholesterol; mood; anxiety; glucose; Triglycerides
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MIND diet (Experimental): The MIND group will consume the MIND diet for 12 weeks.
  Interventions: Other: Mind diet intervention
- MIND plus FB (Experimental): The MIND plus FB intervention will consist of eight sessions.
  Interventions: Other: Mind plus FB intervention
- Usual Care (Other): The routine care group will be instructed to perform daily activities as usual
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Mind diet intervention — These participants will receive four nutrition information sessions, 60 minutes per session, on four consecutive weekdays at the participating community centre. A 7-day sample menu will be developed and explained to the participants as a reference. A nutritionist with the help of a research assistant will conduct each session. The nutritionist-to-participant ratio for each session will be 1:10, 1:11 or 1:12. The following topics will be covered: (1) overview of the MIND diet; (2) discussion with the participants about their ability, motivation and opportunity to adopt the MIND diet; and (3) instruction on how to adopt the MIND diet and how to fill out a logbook for adherence checks.
  Arms: MIND diet
Other: Mind plus FB intervention — The sessions will include four nutritional sessions about the MIND diet and four FB sessions. The participants will be instructed on the MIND diet as previously mentioned. In addition, the MIND-FB participants will undertake four 2 h FB sessions in a country park on four consecutive weekends during daytime hours. The FB sessions will take place during the day if it is sunny, cloudy or lightly raining. The distance covered on each forest visit will be 1-2 kilometres. If it is raining heavily, the session will be cancelled. The participants will gather at the entrance of the country park on the day of FB. The participants will gather at the entrance of the country park on the day of FB. An FB coach will brief the participants and begin the forest trip with a set of experiences on the forest environment. The participants will also be instructed to self-practice FB for 2h per session at weeks 8 & 12 of the intervention.
  Arms: MIND plus FB
Other: Usual care — Participants will receive a health talk and be given pamphlets provided by the Department of Health and/or Hospital Authority about the protective factors and risk factors of CVDs.
  Arms: Usual Care

SUMMARY:
This randomized controlled trial aims to study the effects of the Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) diet combined with forest bathing (FB) on reducing cardiovascular disease (CVD) risk factors in Chinese adults aged 50-75 years at increased risk of CVDs. The study will assess the impact of the intervention on obesity, higher cholesterol, higher blood pressure, higher triglycerides and glucose levels, stress, and negative emotional state.

The investigators hypothesize that the MIND diet combined with FB will have increased cardiac and mental health benefits in Chinese adults with elevated LDL-C compared to the MIND diet alone and routine care. The main questions it aims to answer are:

* What are the effects of the MIND diet plus FB, the MIND diet alone, and routine care on various cardiovascular risk factors and mental health indicators at 4 weeks?
* What is the sustained effect of the MIND diet plus FB, the MIND diet alone, and routine care on these cardiovascular risk factors at 12 weeks?
* How do the effects of the MIND diet plus FB, the MIND diet alone, and routine care differ when considering other individual characteristics such as demographic and lifestyle factors?

This twelve-week study will involve screening participants, obtaining their consent, and measuring various parameters such as blood pressure, lipid panel, glucose levels, waist circumference, body mass index, and dietary intake. Participants will also complete two psychometric questionnaires. Measurements will be taken at three time points: before the intervention, immediately after four weeks of intervention, and at the end of the twelve-week intervention period. Each measurement session is expected to last around 20 minutes.

Participants assigned to the MIND group will attend nutrition group counseling classes and adopt the MIND diet for twelve weeks.

Participants in the MIND plus FB group will attend nutrition group counseling classes and participate in forest bathing sessions.

Participants in the routine-care group will continue their usual activities and receive health talks and pamphlets about cardiovascular diseases.

The investigators will examine and compare the effects of the interventions on cardiovascular risk factors and mental health at 4 weeks and 12 weeks to determine if there are combined and sustained effects.

DETAILED DESCRIPTION:
Background and Significance of the project:

Cardiovascular diseases (CVDs) are the result of atherosclerosis, which is characterized by lipid accumulation and chronic inflammation of the arteries. Elevated low-density lipoprotein cholesterol (LDL-C) is associated with an increased risk of CVDs in all age groups, but particularly in those aged >70 years. The prevalence and burden of CVDs continue to increase globally. In 2019, 523 million people worldwide had a CVD, and CVDs caused 18.6 million deaths and at least 325 million cases of disability. To reduce the risk of developing a CVD, the American College of Cardiology and the American Heart Association have recommended that adults aged 40 to 75 should be prescribed statin therapy if their LDL-C level is >3.4 mmol/L. However, many people are reluctant to initiate statin therapy because they are afraid of potential adverse effects; this reluctance to take statins increases their risk of CVDs and the related morbidity and mortality. Persistent psychosocial stress is a causal risk factor for CVD development. Persistent stress is associated with elevated LDL-C. Recent evidence indicates that adopting a cardioprotective diet in addition to stress management can lower the risk of CVDs .

Stress is widespread in Hong Kong. Owing to their busy lives, many Hong Kong residents consume fast foods, for example, preserved vegetables, processed meat, canned meat, potato crisps and prawn crackers. This unhealthy diet coupled with persistent stress puts people at risk of developing high cholesterol levels and increased blood pressure. The Mediterranean Dietary Approaches to Stop Hypertension (DASH) Intervention for Neurodegenerative Delay (MIND) diet is high in fibre and low in added sugar and is culturally and contextually feasible to adhere to in the metropolis of Hong Kong. The MIND diet encourages increased consumption of plant-based foods, fish, poultry, nuts and berries, which can be easily found in local markets and are accessible and affordable. Adopting the MIND diet has been reported to potentially reduce one's cholesterol level and body weight. Forest bathing (FB) is a relaxation practice in which a person immerses him- or herself in a forest environment to promote physical and mental health. The country parks of Hong Kong are heavily wooded, contain a variety of trees and birds, and are suitable for the practice of FB. FB has been reported to lower blood pressure, anxiety and promoting positive mood but the effect of FB on cardiovascular health benefits is seldom examined in adults. Thus, it is hypothesized that FB could enhance MIND diet on promoting cardiac and mental health. The cardioprotective health benefits of the MIND diet in combination with FB may have an additive effect in reducing CVD risk factors (e.g., LDL-C, blood pressure, stress, BMI, etc.). The investigators conducted a pilot study to examine the combined effect of the MIND diet plus FB in hypertensive adults. The study found that MIND-FB and the MIND diet alone were associated with short-term decreases in LDL-C, blood pressure and anxiety, and they alleviated negative emotions including fatigue, tension-anxiety, confusion and anger among hypertensive adults. The pilot study was conducted among people with hypertension. In the proposed study, the investigators will examine whether the MIND diet combined with FB can also benefit those with high LDL-C. The findings may provide additional preliminary evidence that FB and the MIND diet are therapeutically effective in reducing the CVD risk factors of obesity, high cholesterol and blood pressure, stress and negative emotional states.

This proposed study will target people aged 50-75 years who are at increased risk of CVDs. the investigators will investigate the ability of the MIND diet plus FB to reduce CVD risk factors (obesity, high cholesterol, high blood pressure, high triglycerides and glucose concentrations, stress, and a negative emotional state). The investigators hypothesize that the MIND diet combined with FB will have an increased cardiac and mental health benefit in Chinese adults with elevated LDL-C compared with the MIND diet alone and routine care.

Research plan and methods

Setting and participants: the investigators propose a three-arm randomized controlled trial with a block design (1:1:1) based on the protocols established in our pilot study. Eligible participants will be randomly assigned into three intervention groups: (1) MIND-FB, (2) MIND diet alone and (3) routine care (control). The MIND-FB and MIND groups will receive the intervention, and the control group will receive routine care. Eligible participants will be randomly assigned to one of the three groups by a research assistant based on a predetermined random allocation list generated by a computer program. A serial number will be randomised following block randomisation procedures with a block size of 6 or 12. The participants will be provided with serial numbers, and the research assistant will keep the code for random allocation. The researchers and the data analyst will be blinded to the treatment assignment. The participants will be recruited from the local community through various community centres. An invitation poster will be designed and posted on the website or WhatsApp group of the centres 2 months before the intervention. Potential participants will be required to complete an online demographic questionnaire and undergo health screening to determine eligibility.

Sample size: The pilot study conducted by the project team found that participants in the MIND-FB and MIND groups had a greater benefit in terms of reduced LDL-C than participants who received usual care. For the proposed study, the effect size is estimated to be approximately 0.2. To test a 5% level of significance of the effect among the three groups (MIND-FB, MIND and routine care) on the primary outcome (i.e., reduction in LDL-C at 12 weeks) with a power of 80% and attrition rate of 10% (based on our pilot study), a total of 273 participants will be required. The required sample size will be 91 participants per group (at a ratio of 1:1:1). An F test in G*Power 3.1.9.4 was used to estimate the sample size.

Demographic and other covariates: At the baseline assessment, the investigators will collect sociodemographic data (sex, age, marital status, educational attainment), diet score, physical activity, alcohol consumption, body mass index, waist circumference (cm), self-reported medical diagnoses, measured BP, current medications and number of chronic diseases.

Follow-up during the intervention: A logbook will be given to each participant in the MIND-FB and MIND groups to record their compliance with the MIND diet for adherence checks. A trained research assistant will call the participants every week via WhatsApp to discuss their progress and learning and provide them with feedback if the participant has barriers or challenges in adhering to the MIND diet.

Diet score: Adherence to the MIND dietary pattern will be assessed by calculating the MIND diet score. The MIND diet score assesses 10 healthy food groups and five unhealthy food groups, and a value of 0.0, 0.5 or 1.0 is assigned to each group. In this scoring system, a person receives a score of 1 if they consume items in the healthy food group, while the score is reversed (i.e., -1) for unhealthy food groups. The total MIND diet score is then calculated by summing all food group scores, with a maximum score of 15 representing the strongest adherence to the MIND diet.

Statistical methods: All statistical analyses will be performed using SPSS version 26 (SPSS Inc., Chicago). The alpha level will be set at 0.05 for the two-tailed tests. Intention-to-treat analysis will be applied for any missing data from the follow-ups; multiple imputation will be applied to handle any missing data at baseline. The chi-square test and ANOVA will be used to assess the baseline demographic, socioeconomic and lifestyle characteristics, medical history and medication use among the three groups at baseline. Generalized estimating equation (GEE) models will be used to examine changes in the LDL-C and other secondary outcomes at 4 and 12 weeks and will be adjusted by the random effect of each community centre. Secondary analysis will be conducted to adjust the GEE models for other potential confounders, e.g., demographic characteristics and socioeconomic status. Separate GEE models will be applied to examine dietary changes among the three groups at 4 and 12 weeks.

Ethical considerations: The proposed study will be a health promotion project designed to evaluate the effectiveness of a health promotion activity on cardiac and mental health. Eligible participants will be given an information sheet about the study. Written informed consent will be obtained when the participants are screened for eligibility. The participants will be fully informed about the aims and procedures of the activities and the benefits and risks of participating. The participants will be able to withdraw from the study at any time without consequence. None of the collected data will be revealed to any third party; the data will be kept confidential and anonymous. All data files will be encrypted, and hard copies of the data will be stored in a locked cabinet inside a locked room. The risk of harm to the participants is low. The FB guide and assistant will be first aid providers and will ensure a high level of safety during the FB walk. Individuals with SBP >159 mmHg will be considered ineligible for the study and will be advised to consult a doctor. The contact details of the principal applicant and relevant staff will be provided to the participants in case they have further questions or complaints.

ELIGIBILITY:
Inclusion Criteria:

* age 50-75 years;
* Chinese ethnicity;
* able to speak and understand Cantonese;
* LDL-C point-of-care test (POCT) >2.6 mmol/L;
* State and Trait Anxiety Inventory (STAI) score ≧38;
* physically able to participate in mild-intensity exercise

Exclusion Criteria:

* kidney disease and chronic obstructive pulmonary disease that is poorly controlled,
* known allergies to berries, nuts, fish or olive oil,
* diagnosed mental disorder with medication,
* pregnant,
* those who participated in any relaxation or dietary programme in the past 3 months and those who anticipate joining such a programme in the near future
* those who are unable to walk independently,
* those SBP is more than 159 mmHg.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the mean Low-density lipoprotein cholesterol (LDL-C) at 12 week | From Baseline to 12 weeks.
  The investigators will measure total cholesterol, LDL-C, HDL-C, triglycerides and glucose with the CardioChek Professional Analyser (PA), Point of Care Test (POCT), which has been certified by the United States Food and Drug Administration and by the Centers for Disease Control and Prevention, Cholesterol Reference Method Laboratory Network. The participants will need to fast for 6-8 hours before the POCT.

SECONDARY OUTCOMES:
Change from baseline in the mean Low-density lipoprotein cholesterol (LDL-C) at 4 weeks | From Baseline to 4 weeks.
  The investigators will measure total cholesterol, LDL-C, HDL-C, triglycerides and glucose with the CardioChek Professional Analyser (PA), Point of Care Test (POCT), which has been certified by the United States Food and Drug Administration and by the Centers for Disease Control and Prevention, Cholesterol Reference Method Laboratory Network. The participants will need to fast for 6-8 hours before the POCT.
Change from baseline in the mean High-density lipoprotein cholesterol (HDL-C) at 4 & 12 weeks | From Baseline to 4 & 12 weeks.
  The investigators will measure total cholesterol, LDL-C, HDL-C, triglycerides and glucose with the CardioChek Professional Analyser (PA), Point of Care Test (POCT), which has been certified by the United States Food and Drug Administration and by the Centers for Disease Control and Prevention, Cholesterol Reference Method Laboratory Network. The participants will need to fast for 6-8 hours before the POCT.
Change from baseline in the mean triglycerides at 4 & 12 week | From Baseline to 4 & 12 weeks.
  The investigators will measure total cholesterol, LDL-C, HDL-C, triglycerides and glucose with the CardioChek Professional Analyser (PA), Point of Care Test (POCT), which has been certified by the United States Food and Drug Administration and by the Centers for Disease Control and Prevention, Cholesterol Reference Method Laboratory Network. The participants will need to fast for 6-8 hours before the POCT.
Change from baseline in the mean glucose at 4 & 12 week | From Baseline to 4 & 12 weeks.
  The investigators will measure total cholesterol, LDL-C, HDL-C, triglycerides and glucose with the CardioChek Professional Analyser (PA), Point of Care Test (POCT), which has been certified by the United States Food and Drug Administration and by the Centers for Disease Control and Prevention, Cholesterol Reference Method Laboratory Network. The participants will need to fast for 6-8 hours before the POCT.
Change from baseline in the mean total cholesterol at 4 & 12 week | From Baseline to 4 & 12 weeks.
  The investigators will measure total cholesterol, LDL-C, HDL-C, triglycerides and glucose with the CardioChek Professional Analyser (PA), Point of Care Test (POCT), which has been certified by the United States Food and Drug Administration and by the Centers for Disease Control and Prevention, Cholesterol Reference Method Laboratory Network. The participants will need to fast for 6-8 hours before the POCT.
Change from baseline in the mean systolic blood pressure at 4 & 12 week | From Baseline to 4 & 12 weeks.
  The participants' systolic blood pressure (SBP) will be measured using a digital automatic device (Omron M6 Comfort HEM-7221-E) for BP measurement. This device fulfils the validation criteria of the European Society of Hypertension International Protocol Revision 2010. The blood pressure will be obtained in a seated position after 5 minutes of rest and will be the average of two measurements.
Change from baseline in the mean waist circumference (cm) at 4 & 12 week | From Baseline to 4 & 12 weeks.
  Waist circumference (cm) will be measured between the lower rib and iliac crest using a tape measure.
Change from baseline in the mean body mass index at 4 & 12 week | From Baseline to 4 & 12 weeks.
  The BMI will be calculated using measurements from a height and weight scale.
Change from baseline in the mean anxiety level at 4 & 12 week | From Baseline to 4 & 12 weeks.
  The anxiety level will be assessed using the Chinese version of State and Trait Anxiety Inventory (C-STAI), which has an alpha coefficient to 0.9. It consists of 40 items, in which 20 items each measure state anxiety and trait anxiety. Both state and trait subscales were assessed using a four-point Likert scale, from 1 for "not at all" to 4 for "very much so" for the trait anxiety factor, and from 1 for "almost never" to 4 for "almost always" for the state anxiety factor. The score ranged between 20 and 80. The higher the score is, the greater the anxiety level. It will take each participant about 5-10 minutes to complete the physiological measurement.
Change from baseline in the mean mood state at 4 & 12 week | From Baseline to 4 & 12 weeks.
  The emotional state will be assessed using the Chinese version of Profile of Mood States Short Form (C-POMS-SF), which has a high alpha coefficient to 0.99. It consists of 30 adjectives measured six dimensions of mood: tension-anxiety, depression-dejection, fatigue-inertia, anger-hostility, confusion-bewilderment, and vigor-activity. Ratings were on a five-point Likert scale ranging from 0 (not at all) to 4 (extremely). The total mood disturbance score was obtained by summing the sores on five scales of tension-anxiety, depression-dejection, anger-hostility, fatigue-inertia, and confusion-bewilderment (a constant of +4 is added to the total score of the confusion-bewilderment scale to eliminate the negative score) and subtracting the score of vigor-activity from the total scores. The higher the score, the higher is the level of mood disturbance (ranged from 4 - 124).It will take each participant about 5 -10 minutes to complete the physiological measurement.

OTHER OUTCOMES:
Change from baseline in the mean MIND diet score at 4 & 12 week | From Baseline to 4 & 12 weeks.
  Diet score: Adherence to the MIND dietary pattern will be assessed by calculating the MIND diet score. The MIND diet score assesses 10 healthy food groups and five unhealthy food groups, and a value of 0.0, 0.5 or 1.0 is assigned to each group. In this scoring system, a person receives a score of 1 if they consume items in the healthy food group, while the score is reversed (i.e., -1) for unhealthy food groups. The total MIND diet score is then calculated by summing all food group scores, with a maximum score of 15 representing the strongest adherence to the MIND diet.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Katherine Yau, Doctoral, Principal Investigator — Tung Wah College
Locations (1):
- 16/F, Ma Kam Chan Memorial Building, 31 Wylie Road, Homantin,, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
I would share all individual participant data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: starting 6 months after publication
Access Criteria: investigators whose proposed research has received Institutional Review Boards (IRB) approval

REFERENCES:
- [Background] Aminianfar A, Hassanzadeh Keshteli A, Esmaillzadeh A, Adibi P. Association between adherence to MIND diet and general and abdominal obesity: a cross-sectional study. Nutr J. 2020 Feb 17;19(1):15. doi: 10.1186/s12937-020-00531-1. PMID 32066452
- [Background] Arnett DK, Blumenthal RS, Albert MA, Buroker AB, Goldberger ZD, Hahn EJ, Himmelfarb CD, Khera A, Lloyd-Jones D, McEvoy JW, Michos ED, Miedema MD, Munoz D, Smith SC Jr, Virani SS, Williams KA Sr, Yeboah J, Ziaeian B. 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Sep 10;140(11):e596-e646. doi: 10.1161/CIR.0000000000000678. Epub 2019 Mar 17. No abstract available. PMID 30879355
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2019 Jun 25;73(24):e285-e350. doi: 10.1016/j.jacc.2018.11.003. Epub 2018 Nov 10. No abstract available. PMID 30423393
- [Background] Katsarou AL, Vryonis MM, Protogerou AD, Alexopoulos EC, Achimastos A, Papadogiannis D, Chrousos GP, Darviri C. Stress management and dietary counseling in hypertensive patients: a pilot study of additional effect. Prim Health Care Res Dev. 2014 Jan;15(1):38-45. doi: 10.1017/S1463423612000679. Epub 2013 Feb 21. PMID 23425517
- [Background] Malekmohammad K, Bezsonov EE, Rafieian-Kopaei M. Role of Lipid Accumulation and Inflammation in Atherosclerosis: Focus on Molecular and Cellular Mechanisms. Front Cardiovasc Med. 2021 Sep 6;8:707529. doi: 10.3389/fcvm.2021.707529. eCollection 2021. PMID 34552965
- [Background] Mortensen MB, Nordestgaard BG. Elevated LDL cholesterol and increased risk of myocardial infarction and atherosclerotic cardiovascular disease in individuals aged 70-100 years: a contemporary primary prevention cohort. Lancet. 2020 Nov 21;396(10263):1644-1652. doi: 10.1016/S0140-6736(20)32233-9. Epub 2020 Nov 10. PMID 33186534
- [Background] Morera LP, Marchiori GN, Medrano LA, Defago MD. Stress, Dietary Patterns and Cardiovascular Disease: A Mini-Review. Front Neurosci. 2019 Nov 12;13:1226. doi: 10.3389/fnins.2019.01226. eCollection 2019. PMID 31780892
- [Background] Morris MC, Tangney CC, Wang Y, Sacks FM, Bennett DA, Aggarwal NT. MIND diet associated with reduced incidence of Alzheimer's disease. Alzheimers Dement. 2015 Sep;11(9):1007-14. doi: 10.1016/j.jalz.2014.11.009. Epub 2015 Feb 11. PMID 25681666
- [Background] Morris MC, Tangney CC, Wang Y, Sacks FM, Barnes LL, Bennett DA, Aggarwal NT. MIND diet slows cognitive decline with aging. Alzheimers Dement. 2015 Sep;11(9):1015-22. doi: 10.1016/j.jalz.2015.04.011. Epub 2015 Jun 15. PMID 26086182
- [Background] Roth GA, Mensah GA, Johnson CO, Addolorato G, Ammirati E, Baddour LM, Barengo NC, Beaton AZ, Benjamin EJ, Benziger CP, Bonny A, Brauer M, Brodmann M, Cahill TJ, Carapetis J, Catapano AL, Chugh SS, Cooper LT, Coresh J, Criqui M, DeCleene N, Eagle KA, Emmons-Bell S, Feigin VL, Fernandez-Sola J, Fowkes G, Gakidou E, Grundy SM, He FJ, Howard G, Hu F, Inker L, Karthikeyan G, Kassebaum N, Koroshetz W, Lavie C, Lloyd-Jones D, Lu HS, Mirijello A, Temesgen AM, Mokdad A, Moran AE, Muntner P, Narula J, Neal B, Ntsekhe M, Moraes de Oliveira G, Otto C, Owolabi M, Pratt M, Rajagopalan S, Reitsma M, Ribeiro ALP, Rigotti N, Rodgers A, Sable C, Shakil S, Sliwa-Hahnle K, Stark B, Sundstrom J, Timpel P, Tleyjeh IM, Valgimigli M, Vos T, Whelton PK, Yacoub M, Zuhlke L, Murray C, Fuster V; GBD-NHLBI-JACC Global Burden of Cardiovascular Diseases Writing Group. Global Burden of Cardiovascular Diseases and Risk Factors, 1990-2019: Update From the GBD 2019 Study. J Am Coll Cardiol. 2020 Dec 22;76(25):2982-3021. doi: 10.1016/j.jacc.2020.11.010. PMID 33309175
- [Background] Szczepanska E, Bialek-Dratwa A, Janota B, Kowalski O. Dietary Therapy in Prevention of Cardiovascular Disease (CVD)-Tradition or Modernity? A Review of the Latest Approaches to Nutrition in CVD. Nutrients. 2022 Jun 27;14(13):2649. doi: 10.3390/nu14132649. PMID 35807830
- [Background] Yau KK, Loke AY. Effects of forest bathing on pre-hypertensive and hypertensive adults: a review of the literature. Environ Health Prev Med. 2020 Jun 22;25(1):23. doi: 10.1186/s12199-020-00856-7. PMID 32571202
- [Background] Yau KY, Law PS, Wong CN. Cardiac and Mental Benefits of Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Diet plus Forest Bathing (FB) versus MIND Diet among Older Chinese Adults: A Randomized Controlled Pilot Study. Int J Environ Res Public Health. 2022 Nov 8;19(22):14665. doi: 10.3390/ijerph192214665. PMID 36429384
- [Background] Vale S. Psychosocial stress and cardiovascular diseases. Postgrad Med J. 2005 Jul;81(957):429-35. doi: 10.1136/pgmj.2004.028977. PMID 15998817
- [Background] Shek DT. The Chinese version of the State-Trait Anxiety Inventory: its relationship to different measures of psychological well-being. J Clin Psychol. 1993 May;49(3):349-58. doi: 10.1002/1097-4679(199305)49:33.0.co;2-j. PMID 8315037
- [Background] Chen KM, Snyder M, Krichbaum K. Translation and equivalence: the Profile of Mood States Short Form in English and Chinese. Int J Nurs Stud. 2002 Aug;39(6):619-24. doi: 10.1016/s0020-7489(01)00068-2. PMID 12100873
- [Background] Bolodeoku J, Pinkney S (2019) Imprecision Evaluation of Self-Monitoring of Blood Cholesterol (SMBC) Handheld Point of Care Testing Devices: Elemark™ and Cardiochek PA. Ann Clin Lab Res Vol.7 No.1:290. doi: 10.21767/2386-5180.100290
- [Background] Topouchian J, Agnoletti D, Blacher J, Youssef A, Chahine MN, Ibanez I, Assemani N, Asmar R. Validation of four devices: Omron M6 Comfort, Omron HEM-7420, Withings BP-800, and Polygreen KP-7670 for home blood pressure measurement according to the European Society of Hypertension International Protocol. Vasc Health Risk Manag. 2014 Jan 16;10:33-44. doi: 10.2147/VHRM.S53968. eCollection 2014. PMID 24476688
- [Background] Chen, K. (2000). The Effects of Tai Chi on the Well-being of Community -dwelling Elders in Taiwan, ProQuest Dissertations and Theses. https://ddc-elib-comtw.ezproxy.lb.polyu.edu.hk/doc/9962998
- [Derived] Law PSQ, Yau KY, Wong DC, Yuen KS, Yu CP, Loke AY. Cardioprotective and mentally protective effects of the Mediterranean-dietary approaches to stop hypertension intervention for neurodegenerative delay diet combined with forest bathing among adults with elevated blood cholesterol: a parallel group randomised controlled study protocol. BMJ Open. 2025 Sep 2;15(9):e107982. doi: 10.1136/bmjopen-2025-107982. PMID 40897495
- See also: Sum L. K. (2018 June 6). One in three young Hongkongers suffers from stress, anxiety or depression, Hong Kong playground association survey shows. South China morning Post. Retrieved 2 April 2019 — https://www.scmp.com/news/hong-kong/health-environment/article/2149403/one-three-young-hongkongers-suffers-stress-anxiety
- See also: The Agriculture, Fisheries and Conservation department. (17 August 2022). HONG KONG: THE FACT- Country Parks and Conservation. — http://www.afcd.gov.hk/english//country/cou_lea/the_facts.html